CLINICAL TRIAL: NCT03156582
Title: Impacts of the α-fetoprotein (AFP) Score in Real Life for Patient Selection for Liver Transplantation (LT) for Hepatocellular Carcinoma (HCC)
Acronym: Impact AFP
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC15.170
Record Dates: First submitted 2017-03-27; First posted 2017-05-17 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: liver transplantation, hepatocellular carcinoma, alpha-foetoproteins, AFP
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- all participants included "Milan criteria " and "AFP score": The first arm is made of liver recipients or dropped off list patients at the time of the Milan criteria (fixed until 2013/06/01 for transplanted patients because mandatory three months reevaluation of patients obliged the various teams to respect the criteria at this time, but until 2013/03/01 for dropped off patients because we did not want to count dropped of because of the AFP score in this arm).
  The second arm is made of liver recipients or dropped off list patients at the time of the AFP score (fixed after 2013/06/01)for transplanted patients and after 2013/03/01 for dropped off patients)
  Interventions: Other: Data collecting

INTERVENTIONS:
Other: Data collecting

SUMMARY:
This is a French multicentric retrospective study on intention-to-treat comparing results of LT for HCC before and after the use of the AFP score. The investigators hypothesis is a better respect of the Biomedicine Agency (the French national transplantation agency) criteria since the general application of this score in March 2013. The aim of this study is to determine if the tumoral characteristics at the time of LT are improved and if it modified the patients'outcome.

DETAILED DESCRIPTION:
Liver transplantation is a widely accepted treatment for HCC as it would eliminate the tumour and cure the underlying liver disease. But the success of liver transplantation depends on the tumour load; patients with extensive disease have very poor outcomes, whereas most patients with small tumours can be curred. This had to be taken into account in the context of worldwide organ shortage.

That is why in 1996 Mazzaferro et al. have reported Milan criteria limiting access to liver transplantation for patients with a single tumor ≤ 5 cm or ≤ 3 tumors ≤ 3 cm without tumor invasion or metastasis.

However, in France, these criteria were not respected in about 30% of cases, because they were considered too restrictive and unadapted, with good overall results. This led to the possibility of new criteria definition. Because the value of alpha-foeto-protein was known as a good predictor of tumor aggressivity, a new score emerged in 2012, integrating blocking α-fetoprotein thresholds while allowing an increased number and size of tumors. After validation of this score, the Biomedicine Agency decided to use this α-fetoprotein score, to make the selection of patients allowed to be transplanted since March 2013.

In this multicentric retrospective comparative study The investigators first want to assess if this new score based on imaging is also respected at the explant analysis. Our secondary outcomes are to compare the amount of dropped out patients because of this score, the rate of tumoral relapse, the overall survival and the disease free survival.

The investigators aim at collecting the data of 562 patients registered for Liver Transplantation for Hepatocellular Carcinoma between 2011/03/01 and 2014/03/01 in 5 centres: Paul Brousse (Paris), Montpellier, Lille, Lyon and Grenoble.

ELIGIBILITY:
Inclusion Criteria:

* patients registered for liver transplantation because of Hepatocellular carcinoma between 2011/03/01 and 2014/03/01 in 5 french hospital : Paul Brousse (Paris), Montpellier, Lille Lyon and Grenoble

Exclusion Criteria:

* Patients with a MELD score superior to 20 (because this rate give them access to liver transplantation sooner than the other patients).
* Patients of Domino's grafts
* patients with non hepatocellular tumors on the explanted liver

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients registred for Liver Transplantation because of an Hepatocellular Carcinoma between 2011/03/01 and 2014/03/01 in 5 French centres: Paul Brousse (Paris), Montpellier, Lille, Lyon and Grenoble.
Sampling Method: Non-Probability Sample
Enrollment: 562 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-04-01 (Actual)

PRIMARY OUTCOMES:
Number of participants whose tumoral characteristics on the liver explant were under the criteria of the AFP score | From date of registration for Liver Transplantation until the date of transplantation, assessed up to three years.
  For participants undergoing transplantation, the investigators calculated their AFP score at the time of LT, according to the last value of alphafoetoprotein rate, the number and the size of tumors on the explant. They compared the number of patients whose tumoral characteristics on the liver explant were under the criteria of the AFP score in the two arms.

SECONDARY OUTCOMES:
Rate of patients dropped off list of LT for HCC | From date of registration on the list until the date of exclusion, assessed up to three years.
  Determining if a patient has been excluded by his Transplantation team because of a tumor beyond the Agence de Biomedecine's criteria and comparing the two arms.
Rate of early tumor recurrence after LT for HCC | Two years after liver transplantation
  Determining in the follow up of patients if they present a liver or extra-hepatic recurrence of HCC at 2 years after LT and comparing the two arms.
Rate of tumor recurrence after LT for HCC | From the date of transplantation until the first documented recurrence, assessed through study completion, an average of three years.
  Determining in the follow up of patients after LT if they present a liver or extra-hepatic recurrence of HCC and comparing the two arms.
Overall survival after LT for HCC | From the date of transplantation until the date of death or the date of the last consultation, assessed through study completion, an average of three years
  Calculating the overall survival according to the last follow up of patients after LT and comparing the two arms.
Progression free survival after LT for HCC | From the date of transplantation until the date of first documented recurrence or the date of the last consultation if no recurrence occurs, assessed through study completion, an average of three years.
  Calculating the progressing free survival according to the time of the eventual relapse after LT and comparing the two arms

CONTACTS AND LOCATIONS:
Overall Officials: Thomas DECAENS, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Decaens T, Roudot-Thoraval F, Bresson-Hadni S, Meyer C, Gugenheim J, Durand F, Bernard PH, Boillot O, Boudjema K, Calmus Y, Hardwigsen J, Ducerf C, Pageaux GP, Dharancy S, Chazouilleres O, Dhumeaux D, Cherqui D, Duvoux C. Impact of pretransplantation transarterial chemoembolization on survival and recurrence after liver transplantation for hepatocellular carcinoma. Liver Transpl. 2005 Jul;11(7):767-775. doi: 10.1002/lt.20418. PMID 15973710
- [Background] Decaens T, Roudot-Thoraval F, Hadni-Bresson S, Meyer C, Gugenheim J, Durand F, Bernard PH, Boillot O, Sulpice L, Calmus Y, Hardwigsen J, Ducerf C, Pageaux GP, Dharancy S, Chazouilleres O, Cherqui D, Duvoux C. Impact of UCSF criteria according to pre- and post-OLT tumor features: analysis of 479 patients listed for HCC with a short waiting time. Liver Transpl. 2006 Dec;12(12):1761-9. doi: 10.1002/lt.20884. PMID 16964590
- [Background] Decaens T, Roudot-Thoraval F, Bresson-Hadni S, Meyer C, Gugenheim J, Durand F, Bernard PH, Boillot O, Compagnon P, Calmus Y, Hardwigsen J, Ducerf C, Pageaux GP, Dharancy S, Chazouilleres O, Cherqui D, Duvoux C. Role of immunosuppression and tumor differentiation in predicting recurrence after liver transplantation for hepatocellular carcinoma: a multicenter study of 412 patients. World J Gastroenterol. 2006 Dec 7;12(45):7319-25. doi: 10.3748/wjg.v12.i45.7319. PMID 17143948
- [Background] Decaens T, Roudot-Thoraval F, Badran H, Wolf P, Durand F, Adam R, Boillot O, Vanlemmens C, Gugenheim J, Dharancy S, Bernard PH, Boudjema K, Calmus Y, Hardwigsen J, Ducerf C, Pageaux GP, Hilleret MN, Chazouilleres O, Cherqui D, Mallat A, Duvoux C. Impact of tumour differentiation to select patients before liver transplantation for hepatocellular carcinoma. Liver Int. 2011 Jul;31(6):792-801. doi: 10.1111/j.1478-3231.2010.02425.x. Epub 2011 Mar 31. PMID 21645209
- [Background] Duvoux C, Roudot-Thoraval F, Decaens T, Pessione F, Badran H, Piardi T, Francoz C, Compagnon P, Vanlemmens C, Dumortier J, Dharancy S, Gugenheim J, Bernard PH, Adam R, Radenne S, Muscari F, Conti F, Hardwigsen J, Pageaux GP, Chazouilleres O, Salame E, Hilleret MN, Lebray P, Abergel A, Debette-Gratien M, Kluger MD, Mallat A, Azoulay D, Cherqui D; Liver Transplantation French Study Group. Liver transplantation for hepatocellular carcinoma: a model including alpha-fetoprotein improves the performance of Milan criteria. Gastroenterology. 2012 Oct;143(4):986-94.e3; quiz e14-5. doi: 10.1053/j.gastro.2012.05.052. Epub 2012 Jun 29. PMID 22750200
- [Derived] Brusset B, Dumortier J, Cherqui D, Pageaux GP, Boleslawski E, Chapron L, Quesada JL, Radenne S, Samuel D, Navarro F, Dharancy S, Decaens T. Liver Transplantation for Hepatocellular Carcinoma: A Real-Life Comparison of Milan Criteria and AFP Model. Cancers (Basel). 2021 May 19;13(10):2480. doi: 10.3390/cancers13102480. PMID 34069594